CLINICAL TRIAL: NCT03915340
Title: Single Dose, Full Replicate, Crossover Comparative Bioavailability Study of Propafenone 300 mg Film-Coated Tablets in Healthy Adult Subjects / Fasting State
Brief Title: Bioequivalence Study of Two Formulations of Propafenone 300 mg Film-coated Tablets in Healthy Adult Volunteers After a Single Oral Dose Administration Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmtechnology LLC (Industry)
Collaborators: Altasciences Company Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PTL-P4-227 (v. 2.0 04/09/2019)
Record Dates: First submitted 2019-04-03; First posted 2019-04-16 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-04

CONDITIONS: Bioequivalence
Keywords: propafenone; bioequivalence; Rytmonorm
MeSH Terms: interventions — Propafenone

STUDY DESIGN:
Intervention Model Description: There will be two sequences in the study: A-B-A-B and B-A-B-A, where A = the test product, B = the reference product (see detailed description of A and B items below).
Who Masked: Outcomes Assessor
Masking Description: The randomization code will not be available to the personnel of the bioanalytical facility until the bioanalytical tables have been finalized and audited by the Quality Assurance (QA) department.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence ABAB (Other): 16 subjects assigned to the sequence ABAB will receive a single 300 mg dose of the test product Propafenone (1 x 300 mg film-coated tablet), marked as A in the sequence, in Periods 1 and 3 and a single 300 mg dose of the reference product Rytmonorm (1 x 300 mg film-coated tablet), marked as B in the sequence, in periods 2 and 4. These treatments will be administered orally with approximately 240 mL of water at ambient temperature, in the morning, following a minimum of 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Propafenone; Drug: Rytmonorm
- Sequence BABA (Other): 16 subjects assigned to the sequence BABA will receive a single 300 mg dose of the reference product Rytmonorm (1 x 300 mg film-coated tablet), marked as B in the sequence, in Periods 1 and 3 and a single 300 mg dose of the test product Propafenone (1 x 300 mg film-coated tablet), marked as A in the sequence, in periods 2 and 4. These treatments will be administered orally with approximately 240 mL of water at ambient temperature, in the morning, following a minimum of 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Propafenone; Drug: Rytmonorm

INTERVENTIONS:
Drug: Propafenone — Propafenone is manufactured by Pharmtechnology LLC, Republic of Belarus. Each tablet contains 300 mg of propafenone hydrochloride.
  Other Names: the test product
Drug: Rytmonorm — Rytmonorm is manufactured by Famar Lyon, France (MAH: Mylan Healthcare GmbH, Germany). Each tablet contains 300 mg of propafenone hydrochloride.
  Other Names: the reference product

SUMMARY:
This bioequivalence study will be conducted in healthy male and female volunteers in order to determine the bioequivalence of two different formulations of propafenone after a single oral dose administration under fasting conditions.

DETAILED DESCRIPTION:
This is a single center, randomized, single dose, laboratory-blinded, 2-treatment, 4-period, 2-sequence, full replicate crossover design, in which 32 healthy adult subjects will receive one of the study treatments during each study period.

The intra-subject variation following a single dose of propafenone appears to be around 36% for maximum observed concentration (Cmax) in plasma and around 34% for cumulative area under the concentration time curve calculated from 0 to time of last observed quantifiable concentration using the linear trapezoidal method (AUC0-T). Statistically, given that the expected Test to Reference ratio of geometric least-squares means (LSmeans) should fall within 95 and 105%, it is estimated that the lowest number of subjects to meet the 80 to 125% bioequivalence range with a statistical a priori power of at least 80% is about 28 in a full replicate design study. Therefore, the inclusion of 32 subjects in a full replicate design should be sufficient to account for the possibility of drop-outs, variations around the estimated intra-subject coefficient of variation (CV) and to conclude in favor of the hypothesis of bioequivalence with sufficient statistical power.

Subject eligibility for this study will be determined at the screening visit and eligible subjects will be admitted to the clinical research unit at least 10 hours prior to drug administration for each study period. Food and fluid intake other than water will be controlled for each confinement period and for all subjects. Water will be provided as needed until 1 hour predose. Water will be allowed beginning 1 hour after the administration of the drug.

A subject who withdraws or is withdrawn during the pretrial evaluations but before receiving the investigational product will not be considered as a drop-out and will not be included in the final database. Standbys should be recruited and available to replace any subject who withdraws prior to the first drug administration. On-study drop-outs will not be replaced.

For each study period, subjects will receive a single 300 mg oral dose of propafenone, under fasting conditions and undergo a 36-hour sample collection. Study participants will be aware they will receive different formulations of the same drug, without being informed which product (Test or Reference) is being administered. A total of 21 blood samples will be collected in each study period for pharmacokinetic (PK) assessments. The time of PK blood sample collection will be calculated relative to the time of treatment administration. The actual time of all PK blood draws will be recorded and reported for all subjects.

Subjects are to be discharged from the clinic after the 24-hour postdose PK sample collection, and following medical approval. However, they may be advised to stay at the clinical site for safety reasons, if judged necessary by the physician in charge. Subjects will return to the clinic for blood collection at 36 hours postdose. The drug administrations in each period will be separated by at least 7 calendar days.

The duration of the clinical portion of this study (excluding the screening period) is expected to be approximately 24 days. The actual overall study duration may vary.

Blood samples for PK determination will be processed, split, stored, and shipped according to the sample processing instructions supplied by the bioanalytical facility. Propafenone plasma concentrations will be measured according to a validated bioanalytical method.

Samples from all subjects who received at least one of the investigational products will be assayed and propafenone plasma levels will be reported. The decision of which subjects will be included in the PK analysis is to be documented by the pharmacokineticist (or delegate) and approved by the sponsor before the start of the sample analysis by the bioanalytical facility. The evaluation of plasma PK parameters will take into account all actual PK sampling times.

For the average bioequivalence (unscaled) approach, the calculation of the within-subject standard deviation (Swr), and the scaled-average-bioequivalence analyses, data from those subjects who have at least one evaluable period of Test product and at least one evaluable period of Reference product will be included in the PK and statistical analysis. An unequal number of subjects per sequence may be used. Concentration data of the remaining subjects will be presented separately.

Subjects who do not complete the sampling schedule of one or more study periods may be included in the PK and statistical analysis and bioequivalence determination for only the PK parameters that are judged not to be affected by the missing sample(s).

Statistical inference of propafenone will be based on a bioequivalence (BE) approach using the following standards:

* Average bioequivalence: The ratio of geometric LSmeans with corresponding 90% confidence interval calculated from the exponential of the difference between the Test and Reference product for the ln-transformed parameters Cmax and AUC0-T should all be within the 80.00 to 125.00% bioequivalence range.
* Scaled-average-bioequivalence: In the event that the Cmax Reference-to-Reference within-subject CV is greater than 30%, that its Test-to-Reference geometric LSmeans ratio is within the bioequivalence range of 80.00-125.00% and the average BE criteria is not met, a scaling approach to the bioequivalence assessment will be used. The 90% confidence interval calculated from the exponential of the difference between the Test and Reference product for the ln-transformed parameter Cmax should be within the widened acceptance criteria using scaled-average-bioequivalence.

The safety population will include all subjects who received at least one dose of one of the investigational products. Safety assessments will include physical examination, vital signs, 12-lead ECG, clinical laboratory tests, and adverse event (AE) monitoring. Additional safety measurements may be performed at the discretion of the investigator for reasons related to subject safety. The safety endpoints are the incidence of AEs, laboratory abnormality assessments, vital signs and ECG findings. Any significant changes will be recorded as adverse events only if they are judged clinically significant by the qualified investigator or delegate.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF)
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Healthy adult male or female volunteer
4. A female volunteer must meet one of the following criteria:

   1. Participant is of childbearing potential and agrees to use one of the accepted contraceptive regimens from at least 28 days prior to the first administration of the study drug, during the study and for at least 30 days after the last dose of the study drug. An acceptable method of contraception includes one of the following:

      * Abstinence from heterosexual intercourse
      * Systemic contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch)
      * Intrauterine device (with or without hormones)
      * Condom with intra-vaginally applied spermicide

      Or
   2. Participant whose partner has had a vasectomy less than 6 months prior to dosing, and agrees to use an additional acceptable method of contraception from the first study drug administration through to at least 30 days after the last dose of the study drug

      Or
   3. Participant is of non-childbearing potential, defined as surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or in a menopausal state (i.e. at least 1 year without menses without an alternative medical condition prior to the first study drug administration)
5. A male volunteer meeting one of the following criteria:

   1. Participant is able to procreate and agrees to use one of the accepted contraceptive regimens and not donate sperm from the first study drug administration to at least 90 days after the last drug administration. An acceptable method of contraception includes one of the following:

      * Abstinence from heterosexual intercourse
      * Male condom with spermicide or male condom with a vaginal spermicide (gel, foam, or suppository)

      Or
   2. Participant is unable to procreate; defined as surgically sterile (i.e. has undergone a vasectomy at least 180 days prior to the first study drug administration)
6. Volunteer aged at least 18 years of age but not older than 45 years
7. Volunteer with a body mass index (BMI) greater than or equal to 18.50 and below 30.00 kg/m2
8. Non- or ex-smoker; an ex-smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study drug administration
9. Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without clinical significance, as determined by an investigator
10. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or electrocardiogram (ECG), as determined by an investigator

Exclusion Criteria:

1. Females who are lactating at screening
2. Females who are pregnant according to the pregnancy test at screening or prior to the first study drug administration
3. Seated pulse rate less than 50 Beats per Minute (bpm) or more than 90 bpm at the screening visit or prior to the first study drug administration
4. History of significant hypersensitivity to propafenone or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
5. Presence of significant gastrointestinal, liver or kidney disease, or any other condition known to interfere with drug absorption, distribution, metabolism or excretion, or known to potentiate or predispose to undesired effects
6. History of significant gastrointestinal, liver or kidney disease that may affect drug bioavailability
7. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
8. Presence of out-of-range cardiac interval (PR < 110 msec, PR > 200 msec, QRS < 60 msec, QRS >110 msec and QTc > 440 msec) on the ECG at screening or other clinically significant ECG abnormalities, unless deemed non-significant by the investigator
9. History of myasthenia gravis
10. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
11. Any clinically significant illness in the 28 days prior to the first study drug administration
12. Use of any prescription drugs (with the exception of hormonal contraceptives or hormone replacement therapy) in the 28 days prior to the first study drug administration, that in the opinion of the investigator would put into question the status of the volunteer as healthy
13. Any history of tuberculosis
14. Positive test result for alcohol and/or drugs of abuse at screening or prior to the first drug administration
15. Positive screening results to HIV Ag/Ab Combo, Hepatitis B surface Antigen (HBsAG (B) (hepatitis B)) or Hepatitis C Virus (HCV (C)) tests
16. Volunteers who have already been included in a previous group for this clinical study
17. Volunteers who took propafenone in the 28 days prior to the first study drug administration
18. Volunteers who took an Investigational Product (IP) in the 28 days prior to the first study drug administration
19. Volunteers who donated 50 mL or more of blood in the 28 days prior to the first study drug administration
20. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the 56 days prior to the first study drug administration

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-03-23 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
Cmax of propafenone in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00 hours after each drug administration
  Maximum observed concentration in plasma
AUC0-T of propafenone in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00 hours after each drug administration
  Cumulative area under the concentration time curve calculated from 0 to time of last observed quantifiable concentration (TLQC) using the linear trapezoidal method

SECONDARY OUTCOMES:
Tmax of propafenone in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00 hours after each drug administration
  Time of maximum observed concentration; if it occurs at more than one time point, Tmax is defined as the first time point with this value
TLQC of propafenone in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00 hours after each drug administration
  Time of last observed quantifiable concentration
AUC0-∞ of propafenone in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00 hours after each drug administration
  Area under the concentration time curve extrapolated to infinity, calculated as AUC0-T + ĈLQC (the predicted concentration at time TLQC) / λZ (apparent elimination rate constant)
Residual area of propafenone in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00 hours after each drug administration
  Extrapolated area (i.e. percentage of AUC0-∞ due to extrapolation from TLQC to infinity)
Time point where the log-linear elimination phase begins (TLIN) of propafenone in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00 hours after each drug administration
  Time point where the log-linear elimination phase begins
λZ of propafenone in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00 hours after each drug administration
  Apparent elimination rate constant, estimated by linear regression of the terminal linear portion of the log concentration versus time curve
Thalf of propafenone in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00 hours after each drug administration
  Terminal elimination half-life, calculated as ln(2)/λZ
Number of treatment-emergent adverse events for the test and the reference products | Up to 23 days (after the first drug administration until the completion of clinical part of the study)
  The safety population will include all subjects who received at least one dose of the test or the reference product. Any significant changes will be recorded as treatment-emergent adverse events only if they are judged clinically significant by the qualified investigator or delegate.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Altasciences Company Inc.
Locations (1):
- Altasciences Company Inc., Mount Royal, Quebec, Canada